CLINICAL TRIAL: NCT00526136
Title: Vernakalant (Oral) Prevention of Atrial Fibrillation Recurrence Post-Conversion Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Responsible Party: Gregory Beatch, Ph.D., Vice President, Scientific Affairs, Cardiome Pharma Corp.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1235-SR-202-AF
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo (b.i.d.)
  Interventions: Drug: Placebo
- 2 (Experimental): Vernakalant (oral), 150 mg (b.i.d.)
  Interventions: Drug: Vernakalant (oral)
- 3 (Experimental): Vernakalant (oral), 300 mg (b.i.d.)
  Interventions: Drug: Vernakalant (oral)
- 4 (Experimental): Vernakalant (oral), 500 mg (b.i.d.)
  Interventions: Drug: Vernakalant (oral)

INTERVENTIONS:
Drug: Placebo
  Arms: 1
Drug: Vernakalant (oral) — Vernakalant (oral), 150 mg (b.i.d.) Vernakalant (oral), 300 mg (b.i.d.) Vernakalant (oral), 500 mg (b.i.d.)
  Other Names: RSD1235-SR
  Arms: 2; 3; 4

SUMMARY:
To evaluate the safety, tolerability and efficacy of 3 doses of vernakalant (oral) (150 mg, 300 mg and 500 mg b.i.d.) administered for up to 90 days in subjects with sustained symptomatic atrial fibrillation (AF duration > 72 hours and < 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Comprehend and sign a written informed consent form, (per local and national regulations, as applicable)
* Be 18 to 85 years of age
* Women must not be pregnant, be non-nursing and if pre-menopausal, must be using an effective form of birth control from time of screening until 3 months after the last dose of medication. Methods of birth control considered to be effective may include hormonal contraception (the pill), an intrauterine device (IUD), condoms in combination with a spermicidal cream, total abstinence or sterilisation. Men should be advised not to conceive a child and are advised to use an effective form of birth control from admission until 3 months after the last dose of study medication
* Have symptomatic AF that has been sustained for greater than 72 hours and less than 6 months duration and is clinically indicated for cardioversion;
* Have adequate anticoagulant therapy for cardioversion in accordance with standard of practice as recommended by ACC/AHA/ESC guidelines (Fuster V. et al, 2006);
* Be haemodynamically stable (100 mmHg < systolic blood pressure < 190 mmHg) at screening and on Day 1 before dosing (while taking rate control drugs, if required). After resting supine for 3 minutes, blood pressures should be measured 3 times in 5 minutes with at least 1 minute between assessments;
* Have a body weight between 45 and 113 kg (99 and 250 lbs).

Exclusion Criteria:

* Have known prolonged QT syndrome or QTcB interval of >0.500 sec as measured at screening on a 12 lead ECG; familial long QT syndrome; previous Torsades de Pointes; ventricular fibrillation; or sustained ventricular tachycardia (VT).
* Have a QRS >0.140 sec;
* Documented previous episodes of second or third-degree atrioventricular block;
* Have clinically significant persistent bradycardia with ventricular rate below 50 beats/min, sick-sinus syndrome or pacemaker;
* Have clinically significant moderate or severe aortic valvular stenosis (gradient >25 mmHg), hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy or constrictive pericarditis;
* Have Class III or Class IV congestive heart failure at screening or admission, or have been hospitalized for heart failure in the previous 6 months;
* Have a myocardial infarction (MI), cardiac surgery, angioplasty, unstable angina or acute coronary syndrome within 30 days prior to entry into the study; h) Have serious pulmonary, hepatic, metabolic, renal (serum creatinine > 2.0 mg/dl), gastrointestinal, central nervous system (CNS) or psychiatric disease, end-stage disease states, or any other disease that could interfere with the conduct or validity of the study or compromise subject safety;
* Have known concurrent temporary secondary causes of AF such as alcohol intoxication, pulmonary embolism, hyperthyroidism, pneumonia, hypoxemia (oxygen saturation < 90% on room air), acute pericarditis, or myocarditis;
* Potassium (K+) <3.5 mmol/L or >5.5 mmol/L or magnesium (Mg2+) below the lower limit of normal (Mg2+< 0.65 mmol/L in subjects 65 years or younger and <0.80 mmol/L in subjects 66 years or older). (Both K+ and Mg2+ should be corrected prior to dosing);
* Have clinical evidence of digoxin toxicity;
* Have received an oral Class I or Class III antiarrhythmic agent (including sotalol) within 3 days of randomisation or oral amiodarone within 4 weeks, or have received intravenous Class I or Class III antiarrhythmic agent or i.v. amiodarone within 24 hours prior to start of dosing;
* Have any other surgical or medical condition that, in the judgment of the clinical Investigator might warrant exclusion or be contraindicated for safety reasons;
* Be concurrently participating in another drug study or have received an investigational drug within 30 days prior to screening;
* Be unable to communicate well with the Investigator and to comply with the requirements of the entire study;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2007-03; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Time to first documented recurrence of symptomatic sustained AF. | Time to first documented recurrence of symptomatic sustained AF within Day 90 of dosing
Safety assessments- Vital signs, safety laboratory assays, ECG parameters, physical examinations, and frequency of adverse events | Safety assessments within Day 120 of dosing

SECONDARY OUTCOMES:
Time to first documented recurrence of symptomatic or asymptomatic sustained AF | Time to first documented recurrence of symptomatic or asymptomatic sustained AF within 90 days of dosing
Time to first documented recurrence of symptomatic AF | Time to first documented recurrence of symptomatic AF within 90 days of dosing
Time to first documented recurrence of symptomatic or asymptomatic AF | Time to first documented recurrence of symptomatic or asymptomatic AF within 90 days of dosing
Proportion of subjects in sinus rhythm on Day 90. | Proportion of subjects in sinus rhythm on Day 90 of dosing
Improvement in AF symptoms as assessed by an AF symptom checklist. | Improvement in AF symptoms as assessed by an AF symptom checklist within Day 90 of dosing
Improvement in QOL as measured by SF-36 | Improvement in QOL as measured by SF-36 within Day 90 of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Beatch, PhD, Study Director — Advanz Pharma
Locations (152):
- Australia (5):
  - Royal Adelaide Hospital, Adelaide
  - Royal Hobart Hospital, Hobart
  - Launceston General Hospital, Launceston
  - Queen Elizabeth Hospital, Woodville
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (4):
  - A. Z. Middelheim, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - U. Z. Gasthuisberg, Leuven
  - Heilig Hart Ziekenhuis, Roeselare
- Bulgaria (9):
  - MHAT - Haskovo, Haskovo
  - UMHAT 'Dr. Georgi Stranski', Pleven
  - MHAT 'Rouse AD', Rousse
  - IV MHAT, Sofia
  - MHAT 'Tzaritza Yoanna', Sofia
  - MI Central Clinical Base - Ministry of Interior, Sofia
  - Military Medical Academy, Sofia
  - MHAT 'Sveta Marina', Varna
  - MMA - Hospital Base for Active Treatment - Varna, Varna
- Croatia (4):
  - General Hospital Zadar, Zadar
  - Clinical Hospital Dubrava, Zagreb
  - General Hospital Sveti Duh, Zagreb
  - University Hospital " Merkur ", Zagreb
- Czechia (11):
  - Nemocnice Jindrichuv Hradec, a.s., Jindřichův Hradec
  - Kromerizska Nemocnice, a.s., Kroměříž
  - Nemocnice Kutna Hora s.r.o., Kutná Hora
  - Fakultni Nemocnice Plzen, Pilsen
  - Vojenska Nemocnice Praha, Prague
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Oblastni Nemocnice Pribram, a.s., Příbram
  - Nemocnice v Semilech, Semily
  - Nemocnice Slany, Slaný
  - Nemocnice Tabor, a.s., Tábor
  - Nemocnice Trebic, p.o., Třebíč
- Denmark (6):
  - Bispebjerg Hospital, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
  - Gentofte Amtssygehus, Hellerup
  - Sygehus Vendsyssel - Hjørring, Hjørring
  - Kolding Sygehus, Kolding
  - Region Sjælland Sygehus øst Køge, Køge
- Estonia (4):
  - Viimsi Hospital, Haabneeme
  - Pärnu Hospital, Pärnu
  - North Estonia Regional Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Germany (3):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik Forschungsgesellschaft mbH, Bad Nauheim
  - Evangelisches Krankenhaus, Witten
- Hungary (11):
  - Magyar Imre Hospital, Ajka
  - Baja City Community Hospital, Baja
  - Nyiro Gyula Hospital, Budapest
  - Péterfy Sándor Hospital, Budapest
  - Szent Istvan Hospital, Budapest
  - Bugat Pal Hospital, Gyöngyös
  - Petz Aladár County Teaching Hospital, Győr
  - Bacs-Kiskun County Hospital, Kecskemét
  - Fejér Megyei Szent György Kórház, Székesfehérvár
  - Hetenyi Geza County Hospital, Szolnok
  - Zala County Hospital, Zalaegerszeg
- Lithuania (3):
  - Kaunas Medical University Hospital, Kaunas
  - Klaipeda Seamen's Hospital, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic, Vilnius
- Netherlands (7):
  - VU Medisch Centrum, Amsterdam
  - Reinier de Graaf Groep, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Martini Ziekenhuis, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Stichting Sint Antonius Ziekenhuis, Nieuwegein
  - Isala Klinieken, Zwolle
- New Zealand (4):
  - North Shore Hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Nelson Hospital, Nelson
- Poland (12):
  - SZZOZ Wielospecjalityczny Szpital Miejski im. Dr. E.Warminsk, Bydgoszcz
  - Szpital Powiatowy, Chrzanów
  - Instytut Kardiologii AMG, Gdansk
  - Szpital Miejski w Gdyni, Gdynia
  - Zaklad Farmakologii i Terapii Monitorowanej z Oddzialem Chor, Lodz
  - SP ZOZ Okregowy Szpital Kolejowy, Lublin
  - Szpital Wojewodzki Nr 2, Rzeszów
  - Klinika Kardiologii PAM, Szczecin
  - Szpital Specjalistyczny, Tarnów
  - III Klinika Chorob Wewnetrznych i Kardiologii, Warsaw
  - Wojskowy Instytut Medyczny, CSK MON, Warsaw
  - Osrodek Chorob Serca, 4Wojskowy Szpital Kliniczny z Poliklin, Wroclaw
- Portugal (3):
  - Hospital Fernando da Fonseca, Amadora
  - Hospital de Santa Marta, Lisbon
  - Centro Hospitalar Vila Nova de Gaia, Vila Nova de Gaia
- Romania (10):
  - Spitalul Clinic Judetean de Urgenta Arad, Arad
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Institutul de Cardiologie C.C. Iliescu, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic de Urgenta Sf. Pantelimon, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf. Spiridon Iasi, Lasi
  - Spitalul Clinic Judetean Oradea, Oradea
  - Spitalul Judetean de Urgenta Ploiesti, Ploieşti
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Russia (12):
  - FSI EMC of the President of RF, b.o. City Hospital #51, Moscow
  - MedCentre of RF President, Central Clinical Hospital, Moscow
  - Moscow City Hospital # 29, Moscow
  - Moscow Medical Academy. City Hospital #20, Moscow
  - Moscow SHI City Clinical Hospital #52, Moscow
  - RMA of Postg. education b.o. Botkin City Clinical Hospital, Moscow
  - Russian Cardiology Research Centre, Moscow
  - War Veteran's Hospital #3, Moscow
  - Pokrovskaya City Hospital, Saint Petersburg
  - St- Petersburg GUZ City Hospital #15, Saint Petersburg
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
  - Yaroslavl State Medical Academy b.o. Clinical Hospital #2, Yaroslavl
- Serbia (7):
  - Clinical Center of Serbia, Belgrade
  - Dedinje Cardiovascular Institute, Belgrade
  - Institute of CV Diseases, Clinical Center of Serbia, Belgrade
  - Institute of Cardiovascular Diseases Sremska Kamenica, Kamenitz
  - Clinical Center for Cardiovascular Diseases, Niška Banja
  - Clinical Center Bezanijska Kosa, Zemun
  - Clinical Center Zemun, Zemun
- National Heart Center, Singapore, Singapore
- Slovakia (6):
  - FNsP Bratislava - Pracovisko Stare Mesto, Bratislava
  - Slovensky Ustav Srdcovocievnych Chorob, Bratislava
  - Vychodoslovensky Ustav Srdcovocievnych Chorob, Košice
  - Fakultna Nemocnica Nitra, Nitra
  - FNsP Nove Zamky, Nové Zámky
  - FNsP J. A. Reimana, Prešov
- South Africa (3):
  - Clinresco Centres (Pty) Ltd, Kempton Park
  - Vergelegen Medi-Clinic, Somerset West
  - Clinical Project Research, Worcester
- Spain (7):
  - Hospital Vall D'Hebron, Barcelona
  - Hosp. Virgen de las Nieves, Granada
  - Clinica Universitaria Puerta de Hierro, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Univ. Tarragona Joan XXIII, Tarragona
- Sweden (3):
  - Universitetssjukhuset Malmö, Malmo
  - Universitetssjukhuset Örebro, Örebro
  - Akademiska Sjukhuset, Uppsala
- Switzerland (4):
  - Universitaetsspital Basel, Basel
  - Kantonsspital Liestal, Liestal
  - Cardio Centro Ticino, Lugano
  - Kantonsspital St. Gallen, Sankt Gallen
- Ukraine (13):
  - Reg.Diag.Center of Dnepr., Dnipro
  - Cent.City Clin.Hosp.#3.Chair of Int.Dis.#2 of Donetsk SMU, Donetsk
  - Donetsk Regional Clinical Hospital, Donetsk
  - City Clinical Hospital #8, Kharkiv
  - City Clinical Hospital #1, Kiev
  - Kiev City Clinical Hospital No 5, Coronary Care Unit, Kiev
  - Kiev Clinical Emergency Care Hospital, Kiev
  - M.D.Strazhesko Institut of Cardiology, Kiev
  - N.D. Strazhesko Institute of Cardiology, Kiev
  - Lugansk First Clinical Multiprofile Hospital #1, cardiology, Luhansk
  - Lviv Reg St Clinical Treat-and-Diagn Cardio. Centre, Lviv
  - City Clinical Hospital #9, Odesa
  - Hospital Therapy Dept #1of Zaporozhye SMU, Zaporizhzhya

REFERENCES:
- [Derived] Torp-Pedersen C, Raev DH, Dickinson G, Butterfield NN, Mangal B, Beatch GN. A randomized, placebo-controlled study of vernakalant (oral) for the prevention of atrial fibrillation recurrence after cardioversion. Circ Arrhythm Electrophysiol. 2011 Oct;4(5):637-43. doi: 10.1161/CIRCEP.111.962340. Epub 2011 Aug 14. PMID 21841207
- See also: Related Info — http://www.cardiome.com